CLINICAL TRIAL: NCT01061788
Title: A Phase I Trial of the IGF-1R Antibody AMG 479 in Combination With Everolimus (RAD001) and Panitumumab in Patients With Advanced Cancer (The RAP Trial)
Brief Title: A Trial of AMG 479, Everolimus (RAD001) and Panitumumab in Patients With Advanced Cancer - QUILT-3.007
Acronym: RAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey Clarke (Other)
Collaborators: NantCell, Inc. (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Clarke, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021317
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Advanced Solid Tumors, Non-small Cell Lung Cancer
Keywords: Phase I; Solid Tumor; AMG 479; Panitumumab; Everolimus; RAD001; Duke; Subjects with refractory advanced solid tumors; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ganitumab; Everolimus; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus, AMG 479, Panitumumab (Experimental): Dose Escalation Cohort #, Subjects, Everolimus, AMG 479
  1. 3-6 subjects, Study drug administered per dose level
  2. 3-6 subjects, Study drug administered per dose level
     Expanded Cohort Subjects, Everolimus, AMG 479 20 subjects, study drug administered per dose level
     Dose Escalation, Cohort #, Subjects, Everolimus, AMG 479, Panitumumab
  3. 3-6 subjects, Study drug administered per dose level
  4. 3-6 subjects, Study drug administered per dose level
  Expanded Cohort Subjects, Everolimus, AMG 479, Panitumumab 20 subjects, Study drug administered per dose level
  NSCLC Cohort Subjects, Everolimus, AMG 479, 20 subjects, Study drug administered per dose level
  Interventions: Drug: AMG 479, Everolimus, Panitumumab

INTERVENTIONS:
Drug: AMG 479, Everolimus, Panitumumab — Dose Escalation Cohort #, Subjects, Everolimus, AMG 479
  1. 3-6 subjects, Study drug administered per dose level
  2. 3-6 subjects, Study drug administered per dose level
     Expanded Cohort Subjects, Everolimus, AMG 479 20 subjects, study drug administered per dose level
     Dose Escalation, Cohort #, Subjects, Everolimus, AMG 479, Panitumumab
  3. 3-6 subjects, Study drug administered per dose level
  4. 3-6 subjects, Study drug administered per dose level
  Expanded Cohort Subjects, Everolimus, AMG 479, Panitumumab 20 subjects, Study drug administered per dose level
  NSCLS Cohort Subjects, Everolimus, AMG 479, 20 subjects, Study drug administered per dose level

SUMMARY:
This open-label, non-randomized, dose escalation phase I biomarker trial of the triplet regimen of AMG 479, everolimus, and panitumumab for subjects with refractory advanced solid tumors is designed to assess the safety and tolerability of this combination as well as preliminary efficacy.

DETAILED DESCRIPTION:
The purpose of this study is to find the safest dose of the drugs AMG 479 and everolimus in combination and then with panitumumab added. This study will consist of two parts. If you are enrolled in Part One of the study, you will receive AMG 479 and everolimus. If you are enrolled in Part Two of the study, you will receive AMG 479, everolimus, and panitumumab. The study will also look at how the drugs work in the body, and will see if there is any effect on your cancer.

The study will have two parts: The first part will be to define the MTD/RPTD of the doublet combination of AMG 479 + everolimus using a standard 3-6 subjects per dose level. Since each agent is known to be well tolerated as monotherapy, we will start with the full dose of AMG 479 and escalate the dose of everolimus. Once the RPTD is established, an additional 20 subjects will be added to confirm the tolerability of this regimen and to allow more detailed biomarker assessment for the effect of each agent alone in the doublet combination. In this biomarker expanded cohort, subjects will start treatment with 2 weeks of AMG 479 monotherapy (a single dose of AMG 479), followed by the combination of AMG 479 + everolimus on day 15.

The second part of the study will assess tolerability of the triplet therapy, with panitumumab added to the RPTD of AMG 479 + everolimus, again using a standard cohort size of 3-6 subjects. Finally, at the recommended phase II dose of the triplet therapy, 20 subjects will be added to an expanded safety and biomarker cohort. In this biomarker expanded cohort, 10 subjects will start treatment with two weeks of AMG 479 monotherapy (a single dose of AMG 479), and 10 subjects will start treatment with two weeks of everolimus monotherapy, with all subjects starting the triplet combination therapy with panitumumab on day 15.

Two sustained complete responses (one > 2 years of complete response, second >8 months of complete response) were seen in subjects with refractory NSCLC (never smokers) enrolled in the doublet regimen. Therefore, an additional 20 subjects with NSCLC, never smokers or non-smokers with ≤ 10 year pack smoking history will be enrolled at MTD/RPTD to further assess safety, tolerability and clinical activity in this specific patient cohort. In this cohort, subjects will start both drugs on cycle 1, day 1.

ABOUT THE STUDY DRUGS:

AMG 479 is an intravenous (I.V., meaning through a vein) medication made from a special type of human protein called antibodies. AMG 479 blocks the activity of another protein called IGF-1R which is important for tumors to grow. Blocking IGFR-1 activity has been shown to slow or kill cancer cells in laboratory studies. AMG 479 is currently being evaluated in clinical research studies in a variety of cancers. AMG 479 is not approved by the U.S. Food and Drug Administration (FDA) for the treatment of cancer and is therefore considered an investigational drug.

Everolimus is a pill that works by blocking the activity of a substance in the body known as mTOR (mammalian target of rapamycin). mTOR is important for helping the growth and survival in normal and cancer cells. Blocking mTOR activity has been shown to slow or kill cancer cells in laboratory studies. Everolimus is currently being evaluated in clinical research studies in a variety of cancers. Everolimus (AfinitorTM) is approved by the FDA for the treatment of advanced renal cell carcinoma (kidney cancer), subependymal giant cell astrocytoma (a type of brain cancer), neuroendocrine tumors originating in the lung or gastrointestinal (GI) tract, and HER2-negative breast cancer. Besides cancer, everolimus also has been tested for its ability to help block the rejection of solid organs transplants (such as liver or kidney transplants). Everolimus is approved for this purpose in Europe but not in the United States.

Panitumumab is another intravenous (I.V.) medication made from a special type of human protein called antibodies. Panitumumab blocks the activity of a protein called EGFr which is also important for tumors to grow. Blocking EGFr activity has been shown to slow or kill cancer cells in laboratory studies. Panitumumab is currently being evaluated in clinical research studies in a variety of cancers. Panitumumab (Vectibix™) is approved by the FDA for the treatment of advanced colorectal cancer following 5'FU, oxaliplatin and irinotecan chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed malignant solid tumor that is refractory to standard therapies, or for which no standard therapies exist. Disease must be measurable by RECIST criteria.

   For the NSCLC expanded cohort only: Only histologically proven adenocarcinoma that is refractory to standard therapies.
2. Age >18 years.
3. Karnofsky Performance Status of 60-100.
4. Life expectancy of at least 3 months.
5. Subjects must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count >/=1,500/μl
   * Platelets >/=100,000/μl
   * Magnesium >/= 1.8 mg/dL
   * Phosphorus >/= 2.3 mg/dL
   * Total bilirubin </= 1.5 X upper limit of normal (ULN)
   * AST(SGOT)/ALT(SGPT) </=2.5 X ULN, </=5 X ULN if known hepatic metastases
   * PT/INR; PTT </= 1.3; <1.3 X ULN
   * Creatinine clearance >/=40 mL/min/m2 by Cockroft-Gault or MDRD equation
   * Hemoglobin >9 g/dL
   * Continuation of erythropoietin products is permitted. Hemoglobin must be stable above 9 g/dL for at least 2 weeks without blood transfusion to maintain hemoglobin level.
   * Fasting blood sugar </= 160 mg/dL
   * Patient may be on diabetic medication to achieve glucose control:

     * Documented fasting blood sugars </= 160 mg/dL
     * Diabetic subjects who have recently had their glycemic control regimens adjusted and have documented fasting blood glucose concentrations ≤ 160 mg/dL may be considered regardless of HgbA1c value, if per investigator discretion the subject is considered to have adequate glycemic function
6. Ability to understand and the willingness to sign a written informed consent document.
7. NSCLS expanded cohort only: Total of 20 never smokers and non-smokers. Never smokers are defined as individuals who have never smoked and non-smokers are defined as individuals with a ≤10 pack year history and have quit >15 years

Exclusion Criteria:

1. Radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 28 days prior to day 1 of study drug.

   For the NSCLC expanded cohort only: Palliative radiation therapy ≤14 days of day 1 of study drug.
2. Active CNS metastases. MRI (or CT) required within 3 months of starting treatment for all tumor types known to commonly metastasize to the brain (i.e. all tumors except pancreas, colorectal, ovarian) and for all patients with CNS symptoms that may represent CNS metastases. Metastases which have been treated with radiotherapy > 2 months prior to start of protocol therapy and are asymptomatic (off steroid therapy for at least 1 month) may be included. Patients must have had normal or stable (if treated, no new lesions) brain imaging (CT or MRI) within the two months prior to day 1 of study drug.

   For the NSCLC expanded cohort only: Radiation ≤ 14 days prior to day 1 of study drug. Subjects must be off steroids for > 14 days prior to day 1 of study drug and anticonvulsants must be discontinued.
3. Inadequately controlled hypertension (defined as systolic blood pressure 140 and/or diastolic blood pressure > 90 mmHg). Initiation of antihypertensive is permitted provided adequate control is documented over at least 1 week prior to day 1 of study drug.
4. Evidence of active bleeding diathesis or coagulopathy. For the NSCLC expanded cohort only: History of "blood tinged" sputum allowed.
5. No warfarin therapy. Low molecular weight heparin anticoagulation is permitted provided that patients have been clinically stable on anti-coagulation for at least 2 weeks prior to day 1 of study drug and meet platelet inclusion criteria. No history of active GI bleeding or other major bleeding within previous 6 months prior to day 1 of study drug.
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of study drug (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study.
7. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 1 of study drug.
8. Serious, non-healing wound, ulcer, or bone fracture.
9. Any prior history of hypertensive crisis or hypertensive encephalopathy.
10. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
11. History of clinically significant vascular disease, including any of the following within 6 months prior to day 1 of study drug: myocardial infarction or unstable angina, percutaneous coronary intervention, bypass grafting, ventricular arrhythmia requiring medication, stroke or transient ischemic attack, symptomatic peripheral arterial disease and/or involvement of great vessels by tumor with or without vascular grafting.
12. Chronic treatment with systemic steroids or another immunosuppressive agent with the following exceptions:

    Intermittent steroids may be used on an as-needed basis (e.g. treatment for chemotherapy-related nausea.) Patients on physiologic replacement doses of steroids due to adrenal insufficiency for any reason may remain on these medications.
13. A known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
14. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g. inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection).
15. Patient unwilling to or unable to comply with the protocol.
16. Medical need for the continuous administration of any drugs which affect CYP3A4 though the use of low dose glucocorticoids (e.g. Dexamethasone </= 4 mg daily or equivalent) for anorexia and /or nausea is permitted.
17. History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis, or any evidence of interstitial lung disease on baseline chest CT scan.

    For the NSCLC expanded cohort only: Scarring from previous radiation therapy or pneumonia allowed.
18. Patients who are pregnant and/or lactating are excluded from this study. (The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be embryo- and feto-toxic. Women of child-bearing potential and men must agree to use two forms of adequate contraception (hormonal or barrier method of birth control; abstinence) prior to day 1 of study drug, the duration of study participation and 6 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician and study PI immediately. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. )
19. Other concurrent severe and/or uncontrolled medical, psychiatric or social conditions that could compromise the safety or compliance of treatment as so judged by treating physician. Examples include but are not limited to:

    History of severely impaired lung function defined as spirometry and DLCO that is </= 50% of the normal predicted value and/or 02 saturation that is </= 88% at rest on room air.

    Uncontrolled diabetes mellitus consistent fasting blood glucose readings > 160 mg/dL or < 50 mg/dL). Use of diabetic medications is permitted.

    Hyperlipidemia (>CTC Grade 2: Total Cholesterol > 300-400; Triglycerides > 2.5 ULN). Use of lipid lowering agents is permitted.

    Other: e.g. severe infection, severe malnutrition, ventricular arrhythmias, known active vasculitis of any cause, tumor invasion of any major blood vessel, severe chronic liver or renal disease, active upper GI tract ulceration.
20. No immunizations with attenuated live vaccines within one week of study entry or during study period.

21 Proteinuria at screening as demonstrated by either urine protein: creatinine (UPC) ratio greater than or equal to 1.0 or 24hr collection greater than 1g/24hr at screening.

22 NSCLC cohort only: Current smoker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
To define the maximal tolerated dose (MTD) and/or recommended phase II dose (RPTD) for the doublet AMG 479 in combination with everolimus in subjects with advanced solid tumors. | 3 years
To define the maximal tolerated dose (MTD) and/or recommended phase II dose (RPTD) for the triplet AMG 479 in combination with everolimus and panitumumab in subjects with advanced solid tumors. | 3 years

SECONDARY OUTCOMES:
To describe the toxicity profile seen with these combinations. | 3 years
To describe any signs of clinical activity, including response rate and progression free survival associated with these regimens. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States